CLINICAL TRIAL: NCT04181437
Title: A Phase I Clinical Trial to Evaluate the Pharmacokinetic Interaction and Safety Between NVP-1203-R1 and NVP-1203-R2 in Healthy Adult Subjects
Brief Title: Pharmacokinetic Interaction and Safety Between NVP-1203-R1 and NVP-1203-R2
Acronym: Navipharm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1203_DDI
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NVP-1203-R1 (Experimental): Drug: NVP-1203-R1
  1 tablet, oral dosing
  Interventions: Drug: NVP-1203-R1
- NVP-1203-R2 (Experimental): Drug: NVP-1203-R2
  1 tablet, oral dosing
  Interventions: Drug: NVP-1203-R2
- NVP-1203-R1 and NVP-1203-R2 (Experimental): Drug: NVP-1203-R1 1 tablet and NVP-1203-R2 1 tablet co-administration(oral dosing)
  Interventions: Drug: NVP-1203-R1 and NVP-1203-R2

INTERVENTIONS:
Drug: NVP-1203-R1 — 1 tablet, Single oral dosing
  Other Names: NVP-1203-R1(A)
  Arms: NVP-1203-R1
Drug: NVP-1203-R2 — 1 tablet, Single oral dosing
  Other Names: NVP-1203-R2(E)
  Arms: NVP-1203-R2
Drug: NVP-1203-R1 and NVP-1203-R2 — NVP-1203-R1,1 tablet and NVP-1203-R2, 1 tablet, co-administration, single oral dosing
  Other Names: NVP-1203-R1(A) and NVP-1203-R2(E)
  Arms: NVP-1203-R1 and NVP-1203-R2

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety between NVP-1203-R1 and NVP-1203-R2

DETAILED DESCRIPTION:
pharmacokinetics and safety between NVP-1203-R1 and NVP-1203-R2

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects who signed informed consent

Exclusion Criteria:

* Subjects has a history of allergy reaction of study drug ingredient
* Subjects participated in another clinical trial within 6 months prior to administration of the study drug
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic interaction | 0hours - 24hours
  Area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Y Ran, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, Dongdeok-ro, South Korea

IPD SHARING:
Plan to Share IPD: No